CLINICAL TRIAL: NCT00723788
Title: Magnetic Resonance Evaluation of Appendicitis in Children Aged 8-18
Brief Title: Magnetic Resonance Imaging (MRI) of Appendicitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Pranav Vyas, Assistant Professor of Radiology and Pediatrics, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CNMC4024
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Appendicitis
Keywords: Appendicitis; Children; Magnetic Resonance Imaging
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Only one arm (Experimental): All patients enrolled will receive an MRI of the abdomen with detailed views of the appendix
  Interventions: Device: MRI of the abdomen

INTERVENTIONS:
Device: MRI of the abdomen — Multiple MRI pulse sequences of the abdomen

SUMMARY:
Study to find out if MRI can diagnose appendicitis in children as well as or better than CT scan and/or ultrasound scan performed at the same time. No additional contrast material or sedation will be used to perform the MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-18 years, referred from emergency department for suspected appendicitis and receiving either CT scan or ultrasound of the abdomen for diagnosis

Exclusion Criteria:

* Failure to pass MRI metal screening. Claustrophobia or need for sedation due to inability to hold still.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2008-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pranav K Vyas, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Hormann M, Paya K, Eibenberger K, Dorffner R, Lang S, Kreuzer S, Metz VM. MR imaging in children with nonperforated acute appendicitis: value of unenhanced MR imaging in sonographically selected cases. AJR Am J Roentgenol. 1998 Aug;171(2):467-70. doi: 10.2214/ajr.171.2.9694477.
- [Background] Hormann M, Puig S, Prokesch SR, Partik B, Helbich TH. MR imaging of the normal appendix in children. Eur Radiol. 2002 Sep;12(9):2313-6. doi: 10.1007/s00330-002-1351-0. Epub 2002 May 9. PMID 12195487
- [Background] Pedrosa I, Levine D, Eyvazzadeh AD, Siewert B, Ngo L, Rofsky NM. MR imaging evaluation of acute appendicitis in pregnancy. Radiology. 2006 Mar;238(3):891-9. doi: 10.1148/radiol.2383050146. PMID 16505393
- [Background] Incesu L, Coskun A, Selcuk MB, Akan H, Sozubir S, Bernay F. Acute appendicitis: MR imaging and sonographic correlation. AJR Am J Roentgenol. 1997 Mar;168(3):669-74. doi: 10.2214/ajr.168.3.9057512.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient referral from Emergency Department for suspected appendicitis with ultrasound and/or CT imaging request (0800 hr - 1700 hr) Patients accrued from Aug 2008 - Apr 2010
Groups:
- MRI of the Abdomen: All patients enrolled will receive an MRI of the abdomen with detailed views of the appendix.
Period: Overall Study
Arm/Group | MRI of the Abdomen
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patient referral from Emergency Department for suspected appendicitis with ultrasound and/or CT imaging request (0800 hr - 1700 hr)
Arm/Group | MRI of the Abdomen
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Sensitivity/Specificity and Accuracy of Appendiceal MRI Comparedsurgical Findings or Clinical Follow-up
Description: Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV)
Time Frame: during diagnostic procedure
Population: All patients received MRI, of those 20 also received US and 9 CT, meaning that 8 patients received all three procedures.
Measure: Number; unit: participants
Groups:
- US of the Abdomen: All patients enrolled received an MRI followed in some cases by ultrasund.
- CT of the Abdomen: All patients enrolled received an MRI followed in some cases by computed tomography.
Arm/Group | MRI of the Abdomen | US of the Abdomen | CT of the Abdomen
Number analyzed (Participants) | 21 | 20 | 9
participants
  Sensitivity | 13 | 17 | 4
  Specificity | 19 | 20 | 7
  PPV | 17 | 20 | 4
  NPV | 16 | 18 | 7

ADVERSE EVENTS:
Time Frame: during MRI procedure
Arm/Group | MRI of the Abdomen
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No